CLINICAL TRIAL: NCT00434746
Title: Ascending Multiple Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ILV-094 Administered IV and One Dose of SC Administered to Healthy Subjects
Brief Title: Study of the Safety, Tolerability, PK, and PD of ILV-094 Administered IV or SC to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist, Wyeth
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3199K1-1102
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
MeSH Terms: interventions — fezakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: ILV-094 — Single, ascending doses of 5, 15, 50, 100, 300, and 600 mg IV or SC dose of ILV-094 or placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ascending single IV doses of ILV-094 (an investigational drug) and one SC dose of ILV-094 in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, inpatient/outpatient, sequential-group study of ascending single IV doses of ILV-094 administered to healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 45 years inclusive at screening.
* Body mass index in the range of 17.6 to 26.4 kg/m2 and body weight>45.
* Nonsmoker or smoker of fewer than 10 cigarettes per day. Must be abstain from smoking during inpatient stay.
* Healthy as determined by the investigator on the basis of screening evaluation.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To provide safety, tolerability, PK and immunogenicity profiles | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Ikebukuro, Tokyo, Japan